CLINICAL TRIAL: NCT07211672
Title: Effictiveness of Multichannel Functionnal Electrical Motor and Sensorimotor Stimulation for Subchronic Stroke Gait Rehabilitation
Brief Title: Clinical Implementation of Multichannel Functional Electrical Stimulation Device for Gait Rehabilitation in Subchronic Stroke: A Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Kurage SAS (Other); Natural Sciences and Engineering Research Council, Canada (Other); Clinique Synapse - Réadaptation & Vie Active (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD-25-0532
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stroke Sequelae; Stroke ( 3 Months After Onset)
Keywords: Subchronic stroke; Gait; Rehabilitation; Functionnal electrical stimulation; Motor; Sensorimotor; Multichannel
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multichannel functionnal electrical stimulation (Experimental): The participants will complete 24 rehabilitation sessions over the course of 8 to 12 weeks. During each rehab session, they will receive functionnal electrical stimulation only on their paretic side, the non-paretic side will not receive functionnal electrical stimulation.
  Interventions: Device: Multichannel functionnal electrical stimulation

INTERVENTIONS:
Device: Multichannel functionnal electrical stimulation — The participants completed 24 gait rehabilitation sessions over the course of 8 to 12 weeks. Each session lasted between 30 minutes and 1 hour. A minimum of 2 days seperated two consecutive sessions. The number of sessions was used for standardization of the protocol instead of duration of treatment.
  Four evaluations were completed throughout the protocol. Baseline evaluation(V1) was completed between 2 and 7 days before the first rehabilitation session. Intermediate evaluation(V2) was completed between 2 and 7 days after the 12th rehabilitation session, in other words 4 to 6 weeks after the baseline evaluation (V1) . Post-treatment evaluation(V3) was completed between 2 and 7 days after the 24th rehabilitation session, in other words 8 to 12 weeks after the baseline evaluation (V1). Follow-up evaluation(V4) was completed 2 months(60 days) after the 24th rehabilitation session, in other words 16 to 20 weeks after the baseline evaluation (V1).
  Other Names: Neuroskin

SUMMARY:
The goal of this interventional study is to evaluate the effect of multichannel functionnal electrical stimulation for subchronic stroke gait rehabilitation. The main questions it aims to answer are:

* Does this new therapy help improve walking speed?
* Evaluate other aspects of therapeutic effectiveness such as different aspects of walking endurance, mobility, postural instability and autonomy.
* Evaluate physiological aspects of autonomous gait such as spasticity, muscle strength and motor and sensorimotor recovery.
* Evaluate the acceptability of this new therapy and its effect on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* First ischemic stroke or first hemorrhagic supratentorial stroke
* Stroke must be unique
* Stoke event in the last 12 months but no sooner than 6 months (post subchronic stroke phase)
* Able to walk with the support of one person and one or multiple walking aids (new functionnal ambulatory classification equal to 1, 2 or 3)
* Able to tolerate and respond to electrical stimulation(Muscle strength grading level 3 while having the quadriceps stimulated)
* Willing to delay anti-spastic treatments like botulinic toxins and motor blockers until the end of the rehabilitation period included in the protocol

Exclusion Criteria:

* Multiple strokes
* Does not respond sufficiently to electrical stimulation
* Contraindication to electrical stimulation
* Comprehension, psychiatric or cognitive problems that could hamper the protocol
* Bilateral stroke or subtentorial stroke
* Able to walk without the support of one person (new functionnal ambulatory clssification equal to 4 or more)
* Needing help from more than one person to walk (new functionnal ambulatory classification equal to 0)
* Moderate spasticity in one or more lower body muscle groups (Modified Ashworth Scale Score >= 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed at intermediate evaluation | At baseline evaluation and the intermediate evaluation(4 to 6 weeks after baseline)
  Walking speed was evaluated with a 10 meters walking test without any electrical stimulation. Two trials were done for each evaluation, one at comfortable speed and one at maximal speed. This test is done with a flying start, therefore participants are already at said walking speed when the timer begins. The timer stops when they complete the 10 meters distance. The distance is covered in a straight line. For each speed(comfortable and maximal), the measure is calculated using this formula: Change at V2 = Speed at V2(intermediate) - Speed at V1(baseline).
Change in walking speed at post-treatment evaluation | At baseline evaluation and the post-treatment evaluation(8 to 12 weeks after baseline)
  Walking speed was evaluated with a 10 meters walking test. Two trials were done for each evaluation, one at comfortable speed and one at maximal speed. This test is done with a flying start, therefore participants are already at said walking speed when the timer begins. The timer stops when they complete the 10 meters distance. The distance is covered in a straight line. For each speed(comfortable and maximal), the measure is calculated using this formula:
  Change at V3 = Speed at V3(post-treatment) - Speed at V1(baseline).
Change in walking speed at follow-up evaluation | At baseline evaluation and the follow-up evaluation(16 to 20 weeks after baseline)
  Walking speed was evaluated with a 10 meters walking test. Two trials were done for each evaluation, one at comfortable speed and one at maximal speed. This test is done with a flying start, therefore participants are already at said walking speed when the timer begins. The timer stops when they complete the 10 meters distance. The distance is covered in a straight line. For each speed(comfortable and maximal), the measure is calculated using this formula:
  Change at V4 = Speed at V4(follow-up) - Speed at V1(baseline).

SECONDARY OUTCOMES:
Change in walking endurance at intermediate evaluation | At baseline evaluation and the intermediate evaluation(4 to 6 weeks after baseline)
  Walking endurance was evaluated with a 6 minute walking test. Participants begin walking at the start of the timer. When the participant can't continue walking or when the timer stops, whichever comes first, the distance covered is measured. The distance is covered in a rectangle on flat ground so as to reduce deceleration during turns. Participants performed 2 trials, the maximal distance was kept as the score for the evaluation. Questionnaires were performed in between the two trials, which were separated by at least 30 minutes, so the participants could rest. The measure is calculated using this formula:
  Change at V2 = Distance at V2[intermediate] - Distance at V1[baseline]
Change in walking endurance at post-treatment evaluation | At baseline evaluation and the post-treatment evaluation(8 to 12 weeks after baseline)
  Walking endurance was evaluated with a 6 minute walking test. Participants begin walking at the start of the timer. When the participant can't continue walking or when the timer stops, whichever comes first, the distance covered is measured. The distance is covered in a rectangle on flat ground so as to reduce deceleration during turns. Participants performed 2 trials, the maximal distance was kept as the score for the evaluation. Questionnaires were performed in between the two trials, which were separated by at least 30 minutes, so the participants could rest. The measure is calculated using this formula:
  Change at V3 = Distance at V3[post-treatment] - Distance at V1[baseline]
Change in walking endurance at follow-up evaluation | At baseline evaluation and the follow-up evaluation(16 to 20 weeks after baseline)
  Walking endurance was evaluated with a 6 minute walking test. Participants begin walking at the start of the timer. When the participant can't continue walking or when the timer stops, whichever comes first, the distance covered is measured. The distance is covered in a rectangle on flat ground so as to reduce deceleration during turns. Participants performed 2 trials, the maximal distance was kept as the score for the evaluation. Questionnaires were performed in between the two trials, which were separated by at least 30 minutes, so the participants could rest. The measure is calculated using this formula:
  Change at V4 = Distance at V4[follow-up] - Distance at V1[baseline]
Change in muscle spasticity at intermediate evaluation | At baseline evaluation and intermediate evaluation(4 to 6 weeks after baseline)
  Muscle spasticity was assessed with the Modified Ashworth Scale for 7 lower body muscles groups(Hip: flexors, extensors and adductors, Knee: flexors and extensors, Ankle: flexors and evertors). Each side was scored independently. This scale has 6 levels, minimum is 0(no increase in tone), maximum is 5(segment is rigid in flexion or extension). The value for each visit is the sum of all scores(all muscle group on both sides). The measure is calculated using this formula:
  Change at V2 = Spasticity at V2[intermediate] - Spasticity at V1[baseline]
Change in muscle spasticity at post-treatment evaluation | At baseline evaluation and post-treatment evaluation (8 to 12 weeks after baseline)
  Muscle spasticity was assessed with the Modified Ashworth Scale for 7 lower body muscles groups(Hip: flexors, extensors and adductors, Knee: flexors and extensors, Ankle: flexors and evertors). Each side was scored independently. This scale has 6 levels, minimum is 0(no increase in tone), maximum is 5(segment is rigid in flexion or extension). The value for each visit is the sum of all scores(all muscle group on both sides). The measure is calculated using this formula:
  Change at V3 = Spasticity at V3[post-treatment] - Spasticity at V1[baseline]
Change in muscle spasticity at follow-up evaluation | At baseline evaluation and follow-up evaluation (16 to 20 weeks after baseline)
  Muscle spasticity was assessed with the Modified Ashworth Scale for 7 lower body muscles groups(Hip: flexors, extensors and adductors, Knee: flexors and extensors, Ankle: flexors and evertors). Each side was scored independently. This scale has 6 levels, minimum is 0(no increase in tone), maximum is 5(segment is rigid in flexion or extension). The value for each visit is the sum of all scores(all muscle group on both sides). The measure is calculated using this formula:
  Change at V4 = Spasticity at V4[follow-up] - Spasticity at V1[baseline]
Change in muscle strength at intermediate evaluation | At baseline evaluation and intermediate evaluation (4 to 6 weeks after baseline)
  Muscle strength was assessed on both sides for 10 lower body muscle groups with the Medical Research Council scale for muscle strength. Muscle groups were hip flexors, hip extensors, hip abductors, hip adductors, knee flexors, knee extensors, tibialis anterior, triceps surae, tibialis posterior, fibular muscles. This scale has 6 levels, minimum is 0(no visible contraction), maximum is 5(normal muscle strength). The value for each visit is the sum of all scores(all muscle groups on both sides). The measure is calculated using this formula:
  Change at V2 = Strength at V2[intermediate] - Strength at V1[baseline]
Change in muscle strength at post-treatment evaluation | At baseline evaluation and post-treatment evaluation (8 to 12 weeks after baseline)
  Muscle strength was assessed on both sides for 10 lower body muscle groups with the Medical Research Council scale for muscle strength. Muscle groups were hip flexors, hip extensors, hip abductors, hip adductors, knee flexors, knee extensors, tibialis anterior, triceps surae, tibialis posterior, fibular muscles. This scale has 6 levels, minimum is 0(no visible contraction), maximum is 5(normal muscle strength). The value for each visit is the sum of all scores(all muscle groups on both sides). The measure is calculated using this formula:
  Change at V3 = Strength at V3[post-treatment] - Strength at V1[baseline]
Change in muscle strength at follow-up evaluation | At baseline evaluation and follow-up evaluation (16 to 20 weeks after baseline)
  Muscle strength was assessed on both sides for 10 lower body muscle groups with the Medical Research Council scale for muscle strength. Muscle groups were hip flexors, hip extensors, hip abductors, hip adductors, knee flexors, knee extensors, tibialis anterior, triceps surae, tibialis posterior, fibular muscles. This scale has 6 levels, minimum is 0(no visible contraction), maximum is 5(normal muscle strength). The value for each visit is the sum of all scores(all muscle groups on both sides). The measure is calculated using this formula:
  Change at V4 = Strength at V4[follow-up] - Strength at V1[baseline]
Change in ambulation capacity at intermediate evaluation | At baseline evaluation and intermediate evaluation(4 to 6 weeks after baseline)
  The ambulation capacity is evaluated with the modified emory functional ambulation profile(Baer and Wolf, 2001). It is a timed measure of walking under 5 environnemental challenges, the score is the sum of all timed activities. Minimal value is 0, maximal value is infinite. The measure is calculated using this formula: Change at V2 = Score at V2[intermediate] - Score at V1[baseline]
Change in ambulation capacity at post-treatment evaluation | At baseline evaluation and post-treatment evaluation(8 to 12 weeks after baseline)
  The ambulation capacity is evaluated with the modified emory functional ambulation profile(Baer and Wolf, 2001). It is a timed measure of walking under 5 environnemental challenges, the score is the sum of all timed activities. Minimal value is 0, maximal value is infinite. The measure is calculated using this formula: Change at V3 = Score at V3[post-treatment] - Score at V1[baseline]
Change in ambulation capacity at follow-up evaluation | At baseline evaluation and follow-up evaluation(16 to 20 weeks after baseline)
  The ambulation capacity is evaluated with the modified emory functional ambulation profile(Baer and Wolf, 2001). It is a timed measure of walking under 5 environnemental challenges, the score is the sum of all timed activities. Minimal value is 0, maximal value is infinite. The measure is calculated using this formula: Change at V4 = Score at V4[follow-up] - Score at V1[baseline]
Change in health perception at intermediate evaluation | At baseline evaluation and intermediate evaluation(4 to 6 weeks after baseline)
  Health perception was assessed with the EQ-5D-5L developped by EuroQol Research Foundation. This questionnaire as 5 items(mobility, self-care, usual activities, pain/discomfort, anxiety/depression) all of which have 5 levels(minimum: no problems[1], maximum : incapacitity/extreme problems[5]). The EQ-5D index is then calculated according to the country specific formula using the health state data(Canada=EQ-VT v1.0). The EQ VAS is a visual analog scale ranging from 0(worst health you can imagine) to 100(best health you can imagine). The measure is calculated using this formula:
  Change at V2 = Variable at V2[intermediate] - Variable at V1[baseline]
Change in health perception at post-treatment evaluation | At baseline evaluation and post-treatment evaluation(8 to 12 weeks after baseline)
  Health perception was assessed with the EQ-5D-5L developped by EuroQol Research Foundation. This questionnaire as 5 items(mobility, self-care, usual activities, pain/discomfort, anxiety/depression) all of which have 5 levels(minimum: no problems[1], maximum : incapacitity/extreme problems[5]). The EQ-5D index is then calculated according to the country specific formula using the health state data(Canada=EQ-VT v1.0). The EQ VAS is a visual analog scale ranging from 0(worst health you can imagine) to 100(best health you can imagine). The measure is calculated using this formula:
  Change at V3 = Variable at V3[post-treatment] - Variable at V1[baseline]
Change in health perception at follow-up evaluation | At baseline evaluation and follow-up evaluation(16 to 20 weeks after baseline)
  Health perception was assessed with the EQ-5D-5L developped by EuroQol Research Foundation. This questionnaire as 5 items(mobility, self-care, usual activities, pain/discomfort, anxiety/depression) all of which have 5 levels(minimum: no problems[1], maximum : incapacitity/extreme problems[5]). The EQ-5D index is then calculated according to the country specific formula using the health state data(Canada=EQ-VT v1.0). The EQ VAS is a visual analog scale ranging from 0(worst health you can imagine) to 100(best health you can imagine). The measure is calculated using this formula:
  Change at V4 = Variable at V4[follow-up] - Variable at V1[baseline]
Change in satisfaction with the treatment device at intermediate evaluation | At baseline evaluation and intermediate evaluation(4 to 6 weeks after baseline)
  Patient's satisfaction with the treatment device(Neuroskin) was assessed with the french version of Quebec User Evaluation of Satisfaction with Asisistive Technology (QUEST 2.0). This questionnaire has 16 items, each item uses a 5 point Likert scale(minimum: not satisfied at all[1], maximum: very satisfied[5]). Three variables are analysed:
  1. Satisfaction with the technology: Average of 8 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  2. Satisfaction with the services: Average of 4 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  3. Total score: Average of all 12 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  The measure is calculated using this formula:
  Change at V2 = Variable at V2[intermediate] - Variable at V1[baseline]
Change in satisfaction with the treatment device at post-treatment evaluation | At baseline evaluation and post-treatment evaluation(8 to 12 weeks after baseline)
  Patient's satisfaction with the treatment device(Neuroskin) was assessed with the french version of Quebec User Evaluation of Satisfaction with Asisistive Technology (QUEST 2.0). This questionnaire has 16 items, each item uses a 5 point Likert scale(minimum: not satisfied at all[1], maximum: very satisfied[5]). Three variables are analysed:
  1. Satisfaction with the technology: Average of 8 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  2. Satisfaction with the services: Average of 4 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  3. Total score: Average of all 12 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  The measure is calculated using this formula:
  Change at V3 = Variable at V3[post-treatment] - Variable at V1[baseline]
Change in satisfaction with the treatment device at follow-up evaluation | At baseline evaluation and follow-up evaluation(16 to 20 weeks after baseline)
  Patient's satisfaction with the treatment device(Neuroskin) was assessed with the french version of Quebec User Evaluation of Satisfaction with Asisistive Technology (QUEST 2.0). This questionnaire has 16 items, each item uses a 5 point Likert scale(minimum: not satisfied at all[1], maximum: very satisfied[5]). Three variables are analysed:
  1. Satisfaction with the technology: Average of 8 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  2. Satisfaction with the services: Average of 4 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  3. Total score: Average of all 12 items(minimum: not satisfied at all[1], maximum: very satisfied[5]).
  The measure is calculated using this formula:
  Change at V4 = Variable at V4[follow-up] - Variable at V1[baseline]
Change in functional ambulation classification at intermediate evaluation | At baseline evaluation and intermediate evaluation(4 to 6 weeks after baseline)
  The ambulation capacity is evaluated with the New Functional Ambulation Classification(NFAC) Brun, V., et al. "" Annales de readaptation et de medecine physique. Vol. 43. No. 1. Elsevier Science, 2000. This classification uses 9 levels to differentiate the patient's walking performance with or without help. Minimum score is 0(patient cannot walk or need's help from more than one person), maximum score is 8(patient can walk on flat ground and go up and down stairs without lateral support or using the hand railing). The measure is calculated using this formula:
  Change at V2 = Score at V2[intermediate] - Score at V1[baseline]
Change in functional ambulation classification at post-treatment evaluation | At baseline evaluation and post-treatment evaluation(8 to 12 weeks after baseline)
  The ambulation capacity is evaluated with the New Functional Ambulation Classification(NFAC) Brun, V., et al. "" Annales de readaptation et de medecine physique. Vol. 43. No. 1. Elsevier Science, 2000. This classification uses 9 levels to differentiate the patient's walking performance with or without help. Minimum score is 0(patient cannot walk or need's help from more than one person), maximum score is 8(patient can walk on flat ground and go up and down stairs without lateral support or using the hand railing). The measure is calculated using this formula:
  Change at V3 = Score at V3[post-treatment] - Score at V1[baseline]
Change in functional ambulation classification at follow-up evaluation | At baseline evaluation and post-treatment evaluation(16 to 20 weeks after baseline)
  The ambulation capacity is evaluated with the New Functional Ambulation Classification(NFAC) Brun, V., et al. "" Annales de readaptation et de medecine physique. Vol. 43. No. 1. Elsevier Science, 2000. This classification uses 9 levels to differentiate the patient's walking performance with or without help. Minimum score is 0(patient cannot walk or need's help from more than one person), maximum score is 8(patient can walk on flat ground and go up and down stairs without lateral support or using the hand railing). The measure is calculated using this formula:
  Change at V4 = Score at V4[follow-up] - Score at V1[baseline]